CLINICAL TRIAL: NCT06330506
Title: The Effect of Pressure Ulcer Care Package on the Risk of Surgery-Related Pressure Ulcer Development in Patients Undergoing Orthopaedic Surgery
Brief Title: The Effect of Pressure Ulcer Care Package on the Risk of Pressure Ulcer Development
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Sevgi Deniz Dogan, assistant professor, Cukurova University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 123456123456
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care group (Experimental): The pressure ulcer care package to be prepared by the researchers will be implemented
  Interventions: Other: Pressure ulcer prevention pack
- Standard group (No Intervention): Standard maintenance will be applied

INTERVENTIONS:
Other: Pressure ulcer prevention pack — The pressure ulcer prevention package to be prepared by the researchers will be applied
  Arms: Care group

SUMMARY:
This study aimed to determine the effect of pressure ulcer care package use on the risk of pressure ulcer development due to surgery in patients undergoing orthopedic surgery. It was planned as a randomized controlled study. The population of the study will consist of patients who underwent surgery in the Orthopaedics and Traumatology Clinic of Doğubayazıt Dr.Yaşar Eryılmaz State Hospital Hospital Hospital of Ağrı Provincial Health Directorate. The sample of the study will consist of patients who volunteered to participate in the study that meets the inclusion criteria. To obtain research data, the Personal Information Form developed by the researcher in line with the literature, 3S Operating Theatre Pressure Wound Risk Assessment Scale, Pressure Wound Regions and Stages Monitoring Form prepared according to NPUAP (2016) Pressure Wound Staging System Form will be used. Statistical analysis of the data obtained from the study will be performed using the SPSS 25 (Statistical Package of Social Science) package program.

ELIGIBILITY:
Inclusion Criteria:

* Orthopaedics and traumatology department
* Those who have undergone general or spinal anesthesia
* Without any communication problems
* Patients who volunteered to participate in the study

Exclusion Criteria:

* Patients with pre-operative pressure ulcer
* Those who are bedridden
* Patients referred to the intensive care unit after surgery
* Patients who wish to leave the study will be excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pressure ulcer formation | Three days later
  The 'Pressure Ulcer Sites and Stages Follow-up Form' created by the researchers will be used. With this form, pressure ulcer stages and regions of the patients will be monitored.In this Form, pressure wound stages are classified into stages: Stage I, II, III, IV, Unstageable, Deep Tissue, and Mucosal Membrane Pressure Wound.

CONTACTS AND LOCATIONS:
Locations (1):
- Dogubayazit Dr Yasar Eryılmaz State Hospital, Ağrı, Turkey (Türkiye)